CLINICAL TRIAL: NCT06519292
Title: Immune Checkpoint Inhibitor Associated Cardiovascular Adverse Events in Patients With Cancer
Acronym: ITHACA
Status: Recruiting | Type: Observational
Sponsor: Hanneke W. M. van Laarhoven (Other)
Collaborators: Amsterdam UMC (Other)
Responsible Party: Sponsor-Investigator, Hanneke W. M. van Laarhoven, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Other Study IDs: NL82446.018.22
Record Dates: First submitted 2024-07-18; First posted 2024-07-25 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Cardiovascular Diseases; Arterial Thrombosis; Myocardial Infarction; Stroke; Coronary Artery Disease; Atherosclerosis; Cancer
Keywords: immune checkpoint inhibitors; cardiovascular disease; atherosclerosis
MeSH Terms: conditions — Cardiovascular Diseases; Myocardial Infarction; Stroke; Coronary Artery Disease; Atherosclerosis; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, serum and PBMC
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- ICI group: Patients that receive immune checkpoint inhibitors
  Interventions: Diagnostic Test: Coronary computed tomography angiography (CCTA) at baseline; Diagnostic Test: Coronary computed tomography angiography (CCTA) after 1 year
- Non-ICI group: Patients with similar malignancies, who do not receive immune checkpoint inhibitors
  Interventions: Diagnostic Test: Coronary computed tomography angiography (CCTA) at baseline; Diagnostic Test: Coronary computed tomography angiography (CCTA) after 1 year

INTERVENTIONS:
Diagnostic Test: Coronary computed tomography angiography (CCTA) at baseline — Detailed imaging of coronary arteries
Diagnostic Test: Coronary computed tomography angiography (CCTA) after 1 year — Detailed imaging of coronary arteries

SUMMARY:
Immune checkpoint inhibitors (ICI) have revolutionized cancer treatment and are now approved for various types of cancer. The most common side effects of ICI are immune-related adverse events which can affect any organ or system in the body. Recently, concerns have also risen about cardiovascular effects of ICI. Retrospective studies showed an 4-5 times increased risk of developing an arterial thromboembolic event.

The mechanisms driving the ICI-associated risks of arterial thromboembolic events such as myocardial infarction and stroke, are unclear. Since the risk of a thromboembolism appears to be increased already during the first months after initiation of ICI, immune-related hypercoagulability or (autoimmune) antiphospholipid antibodies may play a role, but data to support this are lacking. The longer-term risk of arterial thromboembolism may be predominantly driven by (accelerated) atherosclerosis, a chronic low-grade inflammatory disease of the larger arteries. Therefore, this study evaluates the effect of ICI on progression of coronary non-calcifid plaque volume by using computed tomography angiography (CCTA).

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed diagnosis of the following tumor types, any stage: esophageal, gastric or junction cancer, colorectal cancer, non-small cell lung carcinoma, melanoma, renal cell carcinoma
* Prior to start of new therapy (i.e. immune checkpoint inhibitor, chemotherapy or follow-up in case of esophageal cancer)
* Age ≥ 50 years

Exclusion Criteria:

* ICI therapy in previous 12 months
* Suspected or confirmed viral, fungal, or bacterial infectious disease
* Use of immunosuppressive therapy prior to ICI start
* Estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m2
* Known allergy to iodinated contrast agents
* Atrial fibrillation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult male or female subjects are eligible for study participation if they have a confirmed cancer diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 214 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Non-calcified coronary plaque volume (difference between baseline and follow-up CT) | 1 year

SECONDARY OUTCOMES:
Plaque characteristics (differences between baseline and follow-up) | 1 year
  Difference in plaque characteristics (i.e. fat attenuation index)
Differences in plasma biomarkers (pro-inflammatory markers) between baseline and follow-up | 3 months, 1 year
  Immune cell composition, T cell composition, IL-1b, IL-6, NLRP3, IL-17, TNF-a, IFN-y
Incidence of Arterial thromboembolic event | 1 year, 5 years
  Incidence of Arterial Thromboembolic events, defined as major cardiovascular events (MACE), including nonfatal ischemic stroke, nonfatal myocardial infarction and cardiovascular death

OTHER OUTCOMES:
Venous thromboembolism | 1 year, 5 years

CONTACTS AND LOCATIONS:
Overall Officials: H.W.M. van Laarhoven, Prof. Dr., Principal Investigator — secretariaat.oncologie@amsterdamumc.nl
Locations (1):
- Amsterdam UMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No